CLINICAL TRIAL: NCT05333601
Title: An eHealth Psychosocial Intervention for Caregivers of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Kimberly Canter, Senior Research Scientist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R03CA235002 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eSCCIP (Experimental): The Electronic Surviving Cancer Competently Intervention Program (eSCCIP) is an innovative eHealth intervention that combines cognitive behavioral and family systems therapy to provide parents and caregivers of children with cancer (PCCC) with evidence-based coping skills and psychosocial support focused on the family unit. eSCCIP has three 30-minute, self-directed, online modules which feature a unique mix of original video content and interactive activities, supplemented by three telehealth follow-up sessions. eSCCIP aims to reduce acute distress and symptoms of post-traumatic stress while increasing positive coping self-appraisal and use of cognitive coping skills.
  Interventions: Behavioral: eSCCIP

INTERVENTIONS:
Behavioral: eSCCIP — The Electronic Surviving Cancer Competently Intervention Program (eSCCIP) is an innovative eHealth intervention that combines cognitive behavioral and family systems therapy to provide parents and caregivers of children with cancer (PCCC) with evidence-based coping skills and psychosocial support focused on the family unit. eSCCIP has three 30-minute, self-directed, online modules which feature a unique mix of original video content and interactive activities, supplemented by three telehealth follow-up sessions. eSCCIP aims to reduce acute distress and symptoms of post-traumatic stress while increasing positive coping self-appraisal and use of cognitive coping skills.

SUMMARY:
The psychosocial needs of children with cancer and their families are well-documented in the literature, including the increased risk of parental posttraumatic stress, parental anxiety, and decreased family functioning. There is a critical need to provide evidence-based psychosocial care to parents of children with cancer, although many challenges exist with regard to in-person intervention delivery. eHealth interventions represent an exciting potential opportunity to address many of the barriers to in-person intervention delivery in this population, but are not yet widely utilized in pediatric psychosocial cancer care. eSCCIP is an innovative eHealth intervention for parents of children with cancer, delivered through a combination of self-guided interactive online content and telehealth follow-up with a therapist. eSCCIP aims to decrease symptoms of anxiety, distress, and posttraumatic stress while improving family functioning by delivering evidence-based therapeutic content through a flexible, easily accessible intervention tool. The four self-guided online modules feature a mix of didactic video content, novel multifamily video discussion groups featuring parents of children with cancer, and hands-on interactive activities. Preliminary Think Aloud testing has been completed and led to several rounds of design and functionality improvements. The objective of the proposed study is to establish feasibility and acceptability of eSCCIP in a diverse group of parents of children with cancer. A secondary, exploratory goal is to evaluate preliminary intervention effectiveness for key psychosocial outcomes. Specific Aim 1 is to identify strategies for increasing participant engagement and retention by conducting focus groups with a diverse sample of parents of children with cancer prior to pilot testing. Specific Aim 2 is to demonstrate the feasibility of eSCCIP through pilot testing with a diverse sample of parents of children with cancer. Specific Aim 3 is to evaluate preliminary effectiveness of eSCCIP through pilot testing with parents of children with cancer. The proposed study is an important first step in meeting a critical need for families of children with cancer and collecting data to power a randomized clinical trial to establish clinical efficacy.

DETAILED DESCRIPTION:
The psychosocial needs of children with cancer and their families are well-documented in the literature, including the increased risk of parental posttraumatic stress, parental anxiety, and decreased family functioning. There is a critical need to provide evidence-based psychosocial care to parents of children with cancer, although many challenges exist with regard to in-person intervention delivery. For example, it can be difficult for parents to schedule additional in-person appointments during cancer treatment, and many pediatric cancer centers lack adequately trained psychosocial staff. eHealth interventions represent an exciting potential opportunity to address many of the barriers to in-person intervention delivery in this population, but are not yet widely utilized in pediatric psychosocial cancer care. eSCCIP is an innovative eHealth intervention for parents of children with cancer, delivered through a combination of self-guided interactive online content and telehealth follow-up with a therapist. eSCCIP aims to decrease symptoms of anxiety, distress, and posttraumatic stress while improving family functioning by delivering evidence-based therapeutic content through a flexible, easily accessible intervention tool. The intervention is grounded in principles of cognitive-behavioral and family systems therapy and is adapted from two efficacious in-person interventions for caregivers of children with cancer, the Surviving Cancer Competently Intervention Program (SCCIP) and the Surviving Cancer Competently Intervention Program - Newly Diagnosed (SCCIP-ND). eSSCIP has been rigorously developed over two years through a stakeholder-engaged development process involving close collaboration with parents of children with cancer, content experts in pediatric oncology and eHealth, and web design and development experts. The four self-guided online modules feature a mix of didactic video content, novel multifamily video discussion groups featuring parents of children with cancer, and hands-on interactive activities. Preliminary Think Aloud testing has been completed and led to several rounds of design and functionality improvements. The objective of the proposed study is to establish feasibility and acceptability of eSCCIP in a diverse group of parents of children with cancer. A secondary, exploratory goal is to evaluate preliminary intervention effectiveness for key psychosocial outcomes. Specific Aim 1 is to identify strategies for increasing participant engagement and retention by conducting focus groups with a diverse sample of parents of children with cancer prior to pilot testing. Specific Aim 2 is to demonstrate the feasibility of eSCCIP through pilot testing with a diverse sample of parents of children with cancer. Specific Aim 3 is to evaluate preliminary effectiveness of eSCCIP through pilot testing with parents of children with cancer. The proposed study is an important first step in meeting a critical need for families of children with cancer and collecting data to power a randomized clinical trial to establish clinical efficacy.

ELIGIBILITY:
Inclusion criteria:

* Participants must be the parent or primary caregiver of a child (ages 0 - 18 years old) diagnosed with cancer.
* Participants must be able to speak and read English.
* Participants must have access to the internet through a computer or mobile device (e.g., smartphone, tablet).

Exclusion Criteria:

- Potential participants are ineligible to participate if their child is not expected to live longer than six months from the time of potential recruitment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Canter, PhD, Principal Investigator — Nemours Children's Health
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | eSCCIP
Started | 44
Completed | 31
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Number enrolled
Arm/Group | eSCCIP
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.86 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 25
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44
Number of Participants that Completed Investigator Derived Baseline Questionnaire [Count of Participants; unit: Participants] | 44

OUTCOME MEASURES:

1. Primary Outcome: The eSCCIP Evaluation Questionnaire
Description: The eSCCIP Evaluation Questionnaire is a questionnaire designed to evaluate intervention acceptability, feasibility, and usability. Data is descriptive and examined at the item-level. Each item is scored on a 0-4 Likert scale (Not at all true - Very true). Mean score with standard deviation are reported at the item-level.
Time Frame: Up to 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 30
score on a scale
  The eSCCIP website was easy to use | 3.53 (0.78)
  The eSCCIP website was convenient to use | 3.6 (0.68)
  eSCCIP was interesting. | 3.76 (0.44)
  I like how eSCCIP looked | 3.6 (0.68)
  I was worried about my privacy when using the eSCCIP website. | 0.33 (0.92)
  It was easy to log-in to the eSCCIP website. | 3.73 (0.58)
  The internet was a good method for delivering eSCCIP. | 3.73 (0.52)
  eSCCIP contained a good mix of videos and "hands on" material. | 3.63 (0.72)
  It was easy to complete telehealth follow-up sessions with the telehealth interventionist. | 3.77 (0.63)
  It was convenient to complete telehealth follow-up sessions with the telehealth interventionist. | 3.80 (0.61)
  The telehealth follow-up sessions were an important part of eSCCIP. | 3.83 (0.46)
  There were enough telehealth follow-up sessions in eSCCIP. | 3.62 (0.68)
  eSCCIP was helpful. | 3.90 (0.31)
  I learned something new from participating in eSCCIP. | 3.90 (0.40)
  It was easy for me to understand the information in eSCCIP. | 3.90 (0.31)
  I trusted the information that was presented in eSCCIP. | 3.93 (0.26)
  The topics covered in eSCCIP were relevant to me. | 3.87 (0.43)
  eSCCIP helped me think differently about cancer. | 3.27 (0.94)
  eSCCIP will help me help my child. | 3.43 (0.77)
  I would recommend eSCCIP to other families. | 3.87 (0.35)
  I was satisfied with eSCCIP. | 3.80 (0.55)

2. Secondary Outcome: Distress Thermometer
Description: Single-item indicator of psychosocial distress that is widely used in the oncology. Scores range from 1-10, with higher scores indicating more distress.
Time Frame: Up to 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 31
score on a scale | 4.03 (2.54)

3. Secondary Outcome: Generalized Anxiety Disorder - 7 (GAD-7)
Description: Questionnaire used to assess state anxiety. Total scores range from 0-21, with higher scores indicating increased anxiety symptom severity.
Time Frame: Up to 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 31
score on a scale | 3.81 (3.89)

4. Secondary Outcome: SCORE-15
Description: Questionnaire used to assess various domains of family functioning. The SCORE-15 generates a cumulative score and three subscales: Strengths and Adaptability (range = 5-25), Overwhelmed by Difficulties (range = 0-20), and Disrupted Communication (range = 0-20). The cumulative sum score ranges from 5-65.
  Higher average scores on the 0-4 and 1-5 scales indicate "worse" family functioning on subscales and the cumulative score.
Time Frame: Up to 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 31
score on a scale
  Total score | 14.74 (5.26)
  Disrupted Communication Subscale | 3.03 (2.11)
  Overwhelmed by Difficulties Subscale | 2.26 (2.13)
  Strengths and Adaptability Subscale | 9.45 (3.75)

5. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: Questionnaire used to assess symptoms of Posttraumatic Stress Disorder (PTSD). Items on the PCL-5 are summed, resulting in cumulative scores ranging from 0-80. Additionally, the PCL-5 provides four index scores that parallel the symptom clusters for a DSM-5 PTSD diagnosis. Initial research suggests an overall cutoff score of 31-33 is clinically significant. Higher scores are indicative of "worse" functioning."
  The score range for Subscale B (5 items) is 0-20. The score range for Subscale C (2 items) is 0-8. The score range for Subscale D (7 items) is 0-28. The score range for Subscale E (6 items) is 0-24. Scoring guidance suggests that cumulative scores are most meaningful in terms of a provisional diagnosis of PTSD. Higher subscale scores are indicative of "worse" functioning for the specific symptom cluster assessed on that subscale.
Time Frame: Up to 9 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 31
score on a scale
  PCL-5 sum score | 11.23 (7.76)
  PCL-5 subscale B | 3.07 (3.07)
  PCL-5 subscale C | 1.55 (1.67)
  PCL-5 subscale D | 3.16 (2.87)
  PCL-5 subscale E | 3.45 (2.50)

6. Secondary Outcome: The COVID-19 Exposure and Family Impact Scales (CEFIS)
Description: Added to study battery after development in response to COVID-19 pandemic. Exploratory analysis. The CEFIS has two parts. Part 1 (Exposure) includes the Exposure scale which consists of 25 Yes/No items with a total score of 0 to 25. Higher scores denote more (negative) exposure.
  Part 2 (Impact) includes the Impact and Distress scales. The Impact scale consists of 10 items which use a 4-point Likert scale (values from 1 - 4) rating impact on participant's and family's life. The mean of the 10 items is the total Impact Scale Score. Higher scores denote a more negative impact. The Distress scale consists of 2 items with a 10-point distress scale (values from 1 - 10 for each item). The mean of these two items is the total Distress Scale Score. Higher scores denote more distress from COVID-19. The values below for Impact and Distress are the average participant subscale scores.
Time Frame: Up to 9 weeks.
Population: The CEFIS was added to the measure battery after the measure was created in response to the onset of the COVID-19 pandemic. As such, only the subset of patients who enrolled after the onset of the pandemic were administered the CEFIS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eSCCIP
Number analyzed (Participants) | 21
score on a scale
  CEFIS Exposure | 7.81 (2.80)
  CEFIS Impact | 2.60 (0.62)
  CEFIS Distress | 4.71 (2.27)

ADVERSE EVENTS:
Time Frame: Up to 9 weeks for each participant, from completion of baseline measures to completion of post-intervention measures.
Description: This is psychosocial intervention study.
Arm/Group | eSCCIP
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT05333601/Prot_SAP_000.pdf